CLINICAL TRIAL: NCT05444517
Title: A Randomized Comparison Between Interscalene And Combined Infraclavicular-Anterior Suprascapular Nerve Blocks For Arthroscopic Shoulder Surgery
Brief Title: Interscalene Block Versus Combined Infraclavicular-Anterior Suprascapular Blocks for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Julian Aliste, Associate Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OAIC 1248/22
Record Dates: First submitted 2022-06-28; First posted 2022-07-06 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative; Shoulder Pain; Surgical Procedure, Unspecified; Diaphragmatic Paralysis
Keywords: Postoperative Shoulder Analgesia; Diaphragmatic Paralysis; Alternative Blocks
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain; Respiratory Paralysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene Block (Active Comparator): Patients randomized to receive an interscalene block.
  Interventions: Procedure: Interscalene Block
- Infraclavicular-Anterior Supraescapular Nerve Blocks (Experimental): Patients randomized to receive a combined infraclavicular plus anterior suprascapular nerve blocks.
  Interventions: Procedure: Infraclavicular - Anterior Supraescapular Nerve Blocks

INTERVENTIONS:
Procedure: Interscalene Block — Ultrasound-guided brachial plexus block injecting 20 ml of bupivacaine 0.5% plus epinephrine 5 micrograms per ml in the Interscalene groove.
  Patients will receive dexamethasone 4 mg intravenously and an ultrasound-guided intermediate cervical plexus block (5 ml of bupivacaine 0.5% plus epinephrine 5 micrograms per ml).
  Other Names: Peripheral Nerve Block
  Arms: Interscalene Block
Procedure: Infraclavicular - Anterior Supraescapular Nerve Blocks — Ultrasound-guided combined infraclavicular-anterior suprascapular block of the brachial plexus, injecting 20 ml of bupivacaine 0.5% plus epinephrine 5 micrograms per ml dorsal to the axillary artery in the infraclavicular fossa plus an ultrasound-guided injection of 3 ml of bupivacaine 0.5% plus epinephrine 5 micrograms per ml under the omohyoid muscle. If the anterior suprascapular nerve could not be identified after five minutes of insonation time, an upper trunk block will be carried out with the same amount of local anesthetic.
  Patients will receive dexamethasone 4 mg intravenously and an ultrasound-guided intermediate cervical plexus block (5 ml of bupivacaine 0.5% plus epinephrine 5 micrograms per ml).
  Other Names: Peripheral Nerve Block
  Arms: Infraclavicular-Anterior Supraescapular Nerve Blocks

SUMMARY:
Postoperative analgesia after shoulder surgery remains a challenge in patients with preexisting pulmonary pathology, as interscalene brachial plexus block (ISB), the standard nerve block for shoulder surgery, carries a prohibitive risk of hemidiaphragmatic paralysis (HDP). Although several diaphragm-sparing nerve blocks have been proposed, none seems to offer equivalent analgesia to ISB while avoiding HDP altogether. For instance, even costoclavicular blocks, which initially fulfilled both requirements, were subsequently found to result in a non-negligible 5%-incidence of HDP.

In this randomized trial, the authors set out to compare ISB and combined infraclavicular block-anterior suprascapular nerve blocks (ICB-ASSNB) for patients undergoing arthroscopic shoulder surgery. The authors hypothesized that ICB-ASSNB would provide equivalent postoperative analgesia to ISB 30 minutes after shoulder surgery and therefore designed the current study as an equivalence trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing arthroscopic shoulder surgery
* American Society of Anesthesiologists classification 1-3
* Body mass index between 20 and 35 kg/mt2

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy (assessed by history and physical examination)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* Obstructive or restrictive pulmonary disease (assessed by history and physical examination)
* Renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* Allergy to local anesthetics (LAs)
* Pregnancy
* Prior surgery in the neck or infraclavicular region
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Static pain 30 minutes after arrival in the post anesthesia care unit (PACU) | 30 minutes after PACU arrival
  Pain intensity at rest using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)

SECONDARY OUTCOMES:
Static pain 1 hour after arrival in the PACU | 1 hour after PACU arrival
  Pain intensity at rest using a NRS ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static pain 3 hours after arrival in the PACU | 3 hours after PACU arrival
  Pain intensity at rest using a NRS ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static pain 6 hours after arrival in the PACU | 6 hours after PACU arrival
  Pain intensity at rest using a NRS ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static pain 12 hours after arrival in the PACU | 12 hours after PACU arrival
  Pain intensity at rest using a NRS ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static pain 24 hours after arrival in the PACU | 24 hours after PACU arrival
  Pain intensity at rest using a NRS ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static pain 36 hours after arrival in the PACU | 36 hours after PACU arrival
  Pain intensity at rest using a NRS ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static pain 48 hours after arrival in the PACU | 48 hours after PACU arrival
  Pain intensity at rest using a NRS ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Block performance time | 1 hour before surgery
  Time from skin disinfection until the end of local anesthetic injection
Intensity of pain during block procedure | 1 hour before surgery
  Evaluated with the Numeric Rating Scale for Pain. This scale is graduated from 0 to 10 points. A 0-point score represents the absence of pain, and a 10-points score represents the worst imaginable pain. Patients will be asked to rate their pain verbally with this scale. The blinded assessor will register the score reported.
Incidence of nerve block side effects | 0 minutes after skin disinfection to 30 minutes after the nerve block
  Determined by the presence of paresthesia, local anesthetic systemic toxicity, vascular puncture, Horner syndrome, or hoarseness after the block.
Sensory and motor block score | 30 minutes after the ending time of local anesthetic injection
  The sensorimotor block will be assessed every 5 minutes until 30 minutes after the end of local anesthetic injection using a 14-point composite score that encompasses the sensory functions of the axillary and supraclavicular nerves as well as the motor functions of the axillary, suprascapular, subscapular and lateral pectoral nerves
  Sensation will be assessed with ice in each nerve territory with a 0 to 2 point scale. 0= no block, patients can feel cold; 1= analgesic block, the patient can feel touch but not cold; 2= anesthetic block, the patient cannot feel cold or touch.
  The motor function will be assessed for each nerve with a 0 to 2 points scale where 0= no motor block; 1= paresis; 2= paralysis.
  Successful blocks at 30 minutes correlate with a final score ( sum of all individual sensory and motor scores) of at least 12 points out of 14, with a sensory score of at least 3 points (out of 4 points).
Block onset time | 1 hour before surgery
  Time required to reach a minimal sensorimotor composite score of 12 points out of a maximum of 14 points. The sensorimotor score is described in outcome 12.
Basal diaphragmatic function | 1 hour before surgery
  Diaphragmatic function evaluated before the nerve block
Incidence of hemidiaphragmatic paralysis (HDP) at 30 minutes after interscalene or infraclavicular-suprascapular block | 30 minutes after the ending time of local anesthetic injection
  HDP will be defined as the absence of diaphragmatic motion during normal respiration coupled with absent or (paradoxical) cranial diaphragmatic movement when the patient forcefully sniffs
Incidence of HDP 30 minutes after PACU arrival | 30 minutes after PACU arrival
  HDP will be defined as the absence of diaphragmatic motion during normal respiration coupled with absent or (paradoxical) cranial diaphragmatic movement when the patient forcefully sniffs
Duration of surgery | 4 hours after skin incision
  Time between skin incision and closure (min)
Postoperative opioid related side effects | 48 hours after PACU arrival
  Presence of postoperative nausea, vomiting, pruritus, urinary retention, respiratory depression.
Intraoperative opioid requirements | Intraoperative period
  Total amount of fentanyl required during general anesthesia
Postoperative opioid consumption | 48 hours after PACU arrival
  Total amount of morphine required during the first 48 hours after surgery
Patient satisfaction | 24 hours after PACU arrival
  Patient satisfaction at 24 hours using a 0-10 scale (0 = not satisfied; 10 = very satisfied)
Persistent neurologic deficit | 7 days after surgery
  Presence of persistent sensory or motor postoperative deficit. The patients will be contacted by telephone and inquired about any sensory or motor deficit in the operated extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Julián Aliste, MD, Principal Investigator — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Tran DQ, Elgueta MF, Aliste J, Finlayson RJ. Diaphragm-Sparing Nerve Blocks for Shoulder Surgery. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):32-38. doi: 10.1097/AAP.0000000000000529. PMID 27941477
- [Background] Tran DQ, Layera S, Bravo D, Cristi-Sanchez I, Bermudez L, Aliste J. Diaphragm-sparing nerve blocks for shoulder surgery, revisited. Reg Anesth Pain Med. 2019 Sep 20:rapm-2019-100908. doi: 10.1136/rapm-2019-100908. Online ahead of print. PMID 31541010
- [Background] Aliste J, Bravo D, Layera S, Fernandez D, Jara A, Maccioni C, Infante C, Finlayson RJ, Tran DQ. Randomized comparison between interscalene and costoclavicular blocks for arthroscopic shoulder surgery. Reg Anesth Pain Med. 2019 Jan 11:rapm-2018-100055. doi: 10.1136/rapm-2018-100055. Online ahead of print. PMID 30635497
- [Background] Sivashanmugam T, Maurya I, Kumar N, Karmakar MK. Ipsilateral hemidiaphragmatic paresis after a supraclavicular and costoclavicular brachial plexus block: A randomised observer blinded study. Eur J Anaesthesiol. 2019 Oct;36(10):787-795. doi: 10.1097/EJA.0000000000001069. PMID 31397702
- [Background] Martinez J, Sala-Blanch X, Ramos I, Gomar C. Combined infraclavicular plexus block with suprascapular nerve block for humeral head surgery in a patient with respiratory failure: an alternative approach. Anesthesiology. 2003 Mar;98(3):784-5. doi: 10.1097/00000542-200303000-00031. No abstract available. PMID 12606927
- [Background] Aliste J, Bravo D, Finlayson RJ, Tran DQ. A randomized comparison between interscalene and combined infraclavicular-suprascapular blocks for arthroscopic shoulder surgery. Can J Anaesth. 2018 Mar;65(3):280-287. doi: 10.1007/s12630-017-1048-0. Epub 2017 Dec 19. PMID 29270914
- [Background] Vorster W, Lange CP, Briet RJ, Labuschagne BC, du Toit DF, Muller CJ, de Beer JF. The sensory branch distribution of the suprascapular nerve: an anatomic study. J Shoulder Elbow Surg. 2008 May-Jun;17(3):500-2. doi: 10.1016/j.jse.2007.10.008. Epub 2008 Feb 11. PMID 18262803
- [Background] Ebraheim NA, Whitehead JL, Alla SR, Moral MZ, Castillo S, McCollough AL, Yeasting RA, Liu J. The suprascapular nerve and its articular branch to the acromioclavicular joint: an anatomic study. J Shoulder Elbow Surg. 2011 Mar;20(2):e13-7. doi: 10.1016/j.jse.2010.09.004. Epub 2010 Dec 30. PMID 21194975
- [Background] Musso D, Flohr-Madsen S, Meknas K, Wilsgaard T, Ytrebo LM, Klaastad O. A novel combination of peripheral nerve blocks for arthroscopic shoulder surgery. Acta Anaesthesiol Scand. 2017 Oct;61(9):1192-1202. doi: 10.1111/aas.12948. Epub 2017 Aug 4. PMID 28776638
- [Background] Tran DQ, Dugani S, Finlayson RJ. A randomized comparison between ultrasound-guided and landmark-based superficial cervical plexus block. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):539-43. doi: 10.1097/AAP.0b013e3181faa11c. PMID 20975470
- [Background] Aliste J, Bravo D, Fernandez D, Layera S, Finlayson RJ, Tran DQ. A Randomized Comparison Between Interscalene and Small-Volume Supraclavicular Blocks for Arthroscopic Shoulder Surgery. Reg Anesth Pain Med. 2018 Aug;43(6):590-595. doi: 10.1097/AAP.0000000000000767. PMID 29630033
- [Background] Spence BC, Beach ML, Gallagher JD, Sites BD. Ultrasound-guided interscalene blocks: understanding where to inject the local anaesthetic. Anaesthesia. 2011 Jun;66(6):509-14. doi: 10.1111/j.1365-2044.2011.06712.x. PMID 21568985
- [Background] Franco CD, Williams JM. Ultrasound-Guided Interscalene Block: Reevaluation of the "Stoplight" Sign and Clinical Implications. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):452-9. doi: 10.1097/AAP.0000000000000407. PMID 27203394
- [Background] Tran DQ, Bertini P, Zaouter C, Munoz L, Finlayson RJ. A prospective, randomized comparison between single- and double-injection ultrasound-guided infraclavicular brachial plexus block. Reg Anesth Pain Med. 2010 Jan-Feb;35(1):16-21. doi: 10.1097/AAP.0b013e3181c7717c. PMID 20048654
- [Background] Maikong N, Kantakam P, Sinthubua A, Mahakkanukrauh P, Tran Q, Leurcharusmee P. Cadaveric study investigating the phrenic-sparing volume for anterior suprascapular nerve block. Reg Anesth Pain Med. 2021 Sep;46(9):769-772. doi: 10.1136/rapm-2021-102803. Epub 2021 Jun 3. PMID 34083356
- [Background] Aguirre O, Tobos L, Reina MA, Sala-Blanch X. Upper trunk block: description of a supraclavicular approach of upper trunk at the points of its division. Br J Anaesth. 2016 Dec;117(6):823-824. doi: 10.1093/bja/aew366. No abstract available. PMID 27956682
- [Background] Aliste J, Cristi-Sanchez I, Bermudez L, Layera S, Bravo D, Tran Q. Assessing surgical anesthesia for shoulder surgery. Reg Anesth Pain Med. 2020 Aug;45(8):675-676. doi: 10.1136/rapm-2019-100981. Epub 2019 Dec 31. No abstract available. PMID 31892544
- [Background] Lloyd T, Tang YM, Benson MD, King S. Diaphragmatic paralysis: the use of M mode ultrasound for diagnosis in adults. Spinal Cord. 2006 Aug;44(8):505-8. doi: 10.1038/sj.sc.3101889. Epub 2005 Dec 6. PMID 16331304
- [Background] Tashjian RZ, Deloach J, Porucznik CA, Powell AP. Minimal clinically important differences (MCID) and patient acceptable symptomatic state (PASS) for visual analog scales (VAS) measuring pain in patients treated for rotator cuff disease. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):927-32. doi: 10.1016/j.jse.2009.03.021. Epub 2009 Jun 16. PMID 19535272